CLINICAL TRIAL: NCT00001715
Title: Evaluation of Hematologic Patients - Training Protocol
Brief Title: Evaluation of Patients With Blood Disorders
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 980090; 98-CC-0090
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-08-23

CONDITIONS: Hematologic Disease
Keywords: Consultation; Training; Referral; Fellowship Program; Outpatient; Blood Disorder
MeSH Terms: conditions — Hematologic Diseases

SUMMARY:
The Hematology Service provides hematology consultations for patients at the Clinical Center and participates in the training of hematology fellows. Patients with a broad range of hematologic disorders must be available in order for the senior staff of the Service to maintain clinical expertise and to provide the breadth of experience necessary for the fellowship program. The purpose of this protocol is to meet these needs by allowing the Hematology Service to see patients with a spectrum of hematologic diseases not studied on existing research protocols at the NIH. These patients will be evaluated over the course of several outpatient visits and returned to the care of their referring physicians.This study was developed to evaluate and possibly treat patients with blood disorders. The Hematology Service of the National Institutes of Health is responsible for the care of patients participating in research studies. In addition the Hematology Service also provides consultation for small groups of patients with blood disorders that have not been diagnosed or that may need special testing.

This study will also provide doctors at the NIH the opportunity to learn more about a wide range of blood disorders and conditions. Patients participating in this study will be evaluated over the course of several outpatient visits and will continue to be cared for by their regular physician.

DETAILED DESCRIPTION:
The Hematology Service provides hematology consultations for patients at the Clinical Center and participates in the training of hematology fellows. Patients with a broad range of hematologic disorders must be available in order for the senior staff of the Service to maintain clinical expertise and to provide the breadth of experience necessary for the fellowship program. The purpose of this protocol is to meet these needs by allowing the Hematology Service to see patients with a spectrum of hematologic diseases not studied on existing research protocols at the NIH. These patients will be evaluated over the course of several outpatient visits and returned to the care of their referring physicians.

ELIGIBILITY:
* INCLUSION CRITERIA:

The patient must have or be suspected of having a blood disorder.

The patient must be clinically stable enough for outpatient evaluation.

The patients must be referred from a physician outside the NIH who will continue to provide the patient's primary medical care.

EXCLUSION CRITERIA:

Inability of patient, parent or legal gaurdian to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 898 (Actual)
Dates: Start 1998-04-21; Study Completion 2017-08-23

CONTACTS AND LOCATIONS:
Overall Officials: Jay N Lozier, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Karalliedde J, Maltese G, Hill B, Viberti G, Gnudi L. Effect of renin-angiotensin system blockade on soluble Klotho in patients with type 2 diabetes, systolic hypertension, and albuminuria. Clin J Am Soc Nephrol. 2013 Nov;8(11):1899-905. doi: 10.2215/CJN.02700313. Epub 2013 Aug 8. PMID 23929932